CLINICAL TRIAL: NCT05359224
Title: Low-dose Prasgurel Versus Clopidogrel on the Dual Antiplatelet Regimen for Intracranial Stenting or Flow Diverter Treatment for Unruptured Cerebral Aneurysms: a Multi-center Randomized Controlled Trial
Brief Title: Low Dose Prasugrel vs Clopidogrel for Stenting or Flow Diverter for Unruptured Aneurysm
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other); Gangnam Severance Hospital (Other); Bucheon St. Mary's Hospital (Other); International St. Mary's Hospital (Unknown); Ewha Woman's University Seoul Hospital (Unknown)
Responsible Party: Principal Investigator, Chang Ki Jang, Assistant professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S6700
Record Dates: First submitted 2022-01-09; First posted 2022-05-03 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysm; Clopidogrel; Prasugrel Hydrochloride
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clopidogrel (Active Comparator): Using a randomization program, the test group (203 patients; Aspirin 100 mg + Prasugrel 5 mg) and control group (203 patients; Aspirin 100 mg + Clopidogrel 75 mg) are classified. Prescribe the above drugs according to the assigned group, and take them 5 days before the procedure.
  Interventions: Drug: Clopidogrel group
- prasugrel (Active Comparator): Using a randomization program, the test group (203 patients; Aspirin 100 mg + Prasugrel 5 mg) and control group (203 patients; Aspirin 100 mg + Clopidogrel 75 mg) are classified. Prescribe the above drugs according to the assigned group, and take them 5 days before the procedure.
  Interventions: Drug: Prasugrel group

INTERVENTIONS:
Drug: Prasugrel group — Prescribe the drugs according to the assigned group, and take them 5 days before the procedure. Perform platelet function test (VerifyNow assay; Accumetrics, San Diego, California) one day before the procedure to check the P2Y12 reaction reactivity. And the hyporesponsive group patient is given prasugrel 5mg once. And aspirin 100mg and prasugrel 5mg will be maintained for 30 days.
  Other Names: effient
  Arms: prasugrel
Drug: Clopidogrel group — Prescribe the drugs according to the assigned group, and take them 5 days before the procedure. Perform platelet function test (VerifyNow assay; Accumetrics, San Diego, California) one day before the procedure to check the P2Y12 reaction reactivity. And the hyporesponsive group patient is given pletaal 100mg once. And aspirin 100mg and clopidogrel 75mg mg will be maintained for 30 days.
  Other Names: plavix
  Arms: Clopidogrel

SUMMARY:
Low clopidogrel response has been reported in about 5-44% of the total population, which is associated with an increase in thromboembolism.

Recently prasugrel drug widely accepted as a good option for these patients. The purpose of this study is to compare the safety and usefulness of prasugrel versus clopidogrel in patients who are scheduled to undergo stent or diverter treatment for non-ruptured cerebral aneurysms.

DETAILED DESCRIPTION:
Unruptured intracranial aneurysm (UIA) is a relatively common disease with a prevalence of about 1% of the total population. Widely accepted techniques of neuro-interventional therapy are coil embolization with or without stent deployment and flow diverter insertion. However, these two techniques inevitably had the risk of thromboembolism. For prevention and decrease, dual antiplatelet therapy is commonly used in the clinical field. However, clopidogrel does not produce normal metabolites due to various internal and external factors in the metabolic process in the liver and eventually fails to perform its original role of platelet activity suppression in many situations, called "clopidogrel hyporesponsive". Low clopidogrel response has been reported in about 5-44% of the total population, which is associated with an increase in thromboembolism.

Recently prasugrel drug widely accepted as a good option for these patients. The purpose of this study is to compare the safety and usefulness of prasugrel versus clopidogrel in patients who are scheduled to undergo stent or diverter treatment for non-ruptured cerebral aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* UIAs without any evidence of rupture in intracranial imaging study within the last 6 months
* Planned treatment with coil embolization with stent insertion or flow diverter insertion
* If the patient himself/herself consented to this study

Exclusion Criteria:

* ∙ History of acute ischemic stroke or transient ischemic attack

  * Any intracranial hemorrhage except subarachnoid hemorrhage due to aneurysm rupture within the last 3 months
  * Concurrent treatment other than endovascular procedure (e.g. open craniotomy and microsurgical clipping)
  * Contraindications to iodine contrast agents
  * Already taking antiplatelet drugs or antithrombotic drugs other than aspirin
  * Hypersensitivity to aspirin, prasugrel or clopidogrel
  * Cardiac arrhythmia that should be needed to take anticoagulants
  * Pregnancy or lactating
  * Chronic kidney disease (< GFR 60)
  * Patients with chronic liver disease who have at least over 100 IU/L of either AST/ALT in the liver function test
  * Patients with pathological active bleeding, such as peptic ulcer
  * Patients with genetic problems, such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption because they contain lactose
  * Patients continuously taking non-steroidal anti-inflammatory drugs (NSAIDs) and cyclooxygenase-2 inhibitors
  * Patients requiring concomitant administration of methotrexate 15 mg or more for one week
  * If it is judged difficult to follow up after treatment

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
peri-procedural thromboembolic complications | 30 days
  * thromboembolism detected during the neurointerventional procedure
  * transient ischemic attack or ischemic stroke or death with evidence of infarction on diffusion weighted imaging, which occurs within 30-days after procedure
    * incidence of treatment-thromboembolic, TIA and death events.

SECONDARY OUTCOMES:
thromboembolic safety endpoint | 30days
  * Ischemic stroke on relevant arterial territory within 30days after procedure or any stroke
  * Diffusion restriction lesion detected on post-procedure 7 days MRI
    * incidence of treatment-ischemic stroke on relevant territory and DWI lesion detected.
bleeding safety endpoint | 30days
  major and minor bleeding within 30days after procedure
  :: incidence of treatment-major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ki Jang, Study Director — Yongin severance hospital,Yonsei university college of medicine
Locations (1):
- Yongin Severance hospital, Yonsei university college of medicine, Gyeonggi-do, Yongin-si, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT05359224/Prot_SAP_002.pdf
  • Informed Consent Form (2022-01-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT05359224/ICF_003.pdf